CLINICAL TRIAL: NCT02167802
Title: Construction and Validation of a Tool for Automatic Identification of Care Pathways At Risk of Sub-optimality in the Management of Severe Infections in Children (DIABACT IV)
Acronym: DIABACT IV
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC14_0119
Record Dates: First submitted 2014-05-07; First posted 2014-06-19 (Estimated); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Severe Infection
Keywords: severe infection, pediatrics, sub-optimal care, term care
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Community bacterial infection remains to this day a common cause of morbidity and mortality in children, which preventability is a challenge for clinicians. In a previous work, the investigators found that 76% supported children admitted to the ICU for severe bacterial infection were appraised as suboptimal and significantly associated with an increased risk of death. In this context, the investigators seek to identify indicators of extractable data PMSI and SNIIR -AM associated with a higher risk of suboptimal early taking care of children with severe bacterial infection in order to combine them and use them as a score or decision tree that the investigators will validate data from a national prospective multicenter study including 512 children admitted to the ICU for severe infection. The investigators then propose a score associated with a risk of suboptimality care to evaluate the performance of the healthcare system .

ELIGIBILITY:
Inclusion Criteria for retrospective inclusions:

* All children from 1 month to 15 years and 3 months admitted in pediatric resuscitation;
* Community with severe bacterial infection defined by a bacterial infection documented by the presence of a bacterium from a normally sterile site (pleural cerebrospinal fluid joint fluid, blood, bone biopsy ...), a positive urine culture on a sampling done in aseptic conditions accompanied by a febrile illness (eg pyelonephritis), or purpura fulminans in the absence of documentation.

Inclusion Criteria for prospective inclusions:

* The inclusion criteria DIABACT III will be expanded to include children 0-1 months.
* Parents and patient (if applicable) who signed the consent biocollection for participation in the substudy.

Exclusion Criteria:

* Nosocomial Infections as defined by the Ministry of Health in its January 2007 issue on nosocomial infections namely: Nosocomial infections are infections acquired in a healthcare facility. Infection is considered nosocomial if it was absent at the time of admission of the patient in the health facility. When the infectious status of the patient at admission is unknown, the infection is generally considered nosocomial if it occurs after a period of at least 48 hours of hospitalization or a period longer than the incubation period of the infection. In case of surgical site infection, the period commonly allowed is 30 days, or if it has been set in place a prosthesis or implant, a year after the intervention.
* Children with whooping cough, bronchiolitis or viral infections

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients included in this study will be children admitted to pediatric intensive care unit for a severe bacterial infection community.
  Retrospective inclusions (data DIABACT III study) of children from 1 month to 15 years and 3 months and prospective inclusions concern for children from 0 months to 15 years and 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 524 (Actual)
Dates: Start 2015-03-20 (Actual); Primary Completion 2020-03-07 (Actual); Study Completion 2020-03-07 (Actual)

PRIMARY OUTCOMES:
the optimality of care questionnaire | 1 month
  optimality of care will be assessed by 2 independent experts, blinded to outcome and final diagnosis. Medical charts will be summarized and given to experts without outcome or diagnosis. They would be asked to evaluate optimality of care as follow: optimal, certainly sub-optimal, possibly suboptimal and not evaluable

SECONDARY OUTCOMES:
outcome at the hospital discharge defined as death, survival without sequelae and survival with sequelae | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Christèle Gras Le Guen, Pr, Principal Investigator — Nantes University Hospital
Locations (12):
- France (12):
  - AP-HP, Paris, France
  - Angers University Hospital, Angers
  - Olivier Brissaud, Bordeaux
  - Jacques Sizun, Brest
  - Thierry Debillon, Grenoble
  - Stéphane Leteurtre, Lille
  - Etienne Javouhey, Lyon
  - Gilles Cambonie, Montpellier
  - Elise Launay, Nantes
  - Stéphane Dauger, Paris
  - Sylvain Renolleau, Paris
  - Hugues Patural, Saint-Etienne